CLINICAL TRIAL: NCT01063894
Title: A Randomized, Controlled, Parallel Trial to Evaluate the Effects of Breakfast on Cognitive Processes in Children
Brief Title: Effects of Breakfast on Cognitive Processes in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kellogg Company (Industry)
Collaborators: Provident Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRV-09013
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2015-08

CONDITIONS: Cognitive Function
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- breakfast cereal (Experimental): breakfast cereal and milk
  Interventions: Other: breakfast cereal
- water (Placebo Comparator): water
  Interventions: Other: water

INTERVENTIONS:
Other: breakfast cereal — breakfast cereal and milk
  Arms: breakfast cereal
Other: water — water
  Arms: water

SUMMARY:
The objective of this study is to test the effects of breakfast on cognitive processing ability in children.

DETAILED DESCRIPTION:
Breakfast consumption has previously been shown to positively affect cognitive and academic performance in children. Specifically, breakfast consumption has been reported to improve memory, attention, problem solving, and logical reasoning compared to the absence of breakfast. This has been found under both short-term laboratory conditions and within a school environment in children from both a low and high socioeconomic background, although some studies have failed to find favorable effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to maintain their habitual diet and physical activity patterns throughout the study period
* Provision of assent by subject
* Subject's guardian provides informed consent to participate in the study and authorization for release of relevant protected health information to the study investigators

Exclusion Criteria:

* Diagnosis of attention deficit disorder, with or without hyperactivity
* A diagnosis of diabetes mellitus
* Acute illness or use of antibiotics within 5 days of visit
* Subject is a non-breakfast eater defined as not regularly eating food prior to 1000 h
* Known sensitivity or allergy to any ingredients of the study product
* Use of any psychotropic medication within 4 weeks
* Subject did not previously participate in an earlier trial with the same study products
* Exposure to investigational agent within 30 days.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide assent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 291 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Quality of Memory and Attention based on results using CDR System | 4 hours following breakfast

SECONDARY OUTCOMES:
Speed of Memory and Attention based on results using CDR System | 4 hours following breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, Ph.D., Study Director — Provident Clinical Research
Locations (1):
- Provident Clinical Research, Addison, Illinois, United States